CLINICAL TRIAL: NCT00881270
Title: Safety Dermatological Evaluation: Acceptability With Paediatric Follow up Dermacyd Infantile (Lactic Acid).
Brief Title: Dermacyd Infantile - Acceptability.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04678
Record Dates: First submitted 2009-04-10; First posted 2009-04-15 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Hygiene

ARMS (1):
- Dermacyd infantile (Lactic Acid) (Experimental): treatment duration 21 consecutive days
  Interventions: Drug: LACTIC ACID(ND)

INTERVENTIONS:
Drug: LACTIC ACID(ND) — Dermacyd Infantile (LACTIC ACID)

SUMMARY:
Primary Objective:

To prove the safety of the formulation in normal conditions of use.

ELIGIBILITY:
Inclusion criteria:

* Integral skin test in the region
* Use the same category of cosmetics
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time.

Exclusion criteria:

* Use of Anti-inflammatory, immunosuppressant or anti-histaminic drugs
* Allergic or atopic history to cosmetics products
* Cutaneous active disease (local or general) in the evaluated area
* Disease which can cause immunosuppressant, such as diabetes, HIV
* Endocrine pathology
* Intensive solar exposure until 15 days before evaluation
* Treatment four months before selection.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The absence of irritation and the good acceptability will be evaluated using one specific scale which describes the intensity of the reaction. | From the treatment start to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil